CLINICAL TRIAL: NCT02489058
Title: A Retrospective/Prospective Analysis of Characterization of the Long-Term Responders on Olaparib in Solid Tumours
Brief Title: A Study of Long-Term Responders on Olaparib
Acronym: OLALA
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: OZM-061
Record Dates: First submitted 2015-04-24; First posted 2015-07-02 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — * Archival tumor tissue sample for biomarker research
  * Optional fresh tumor tissue sample for biomarker research (if participants are still on olaparib and their disease progressed)
  * Blood sample for pharmacokinetics (if participants are still on olaparib)
  * Blood sample for pharmacogenomics (if participants are still on olaparib and their disease progressed)
  * Blood samples for circulating tumor DNA (if participants are still on olaparib)
  * Blood sample for germline BRCA1/2 testing if not previously done (if participants are still on olaparib and their disease progressed)
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational and sample collection study involving patients (alive or deceased) from several clinical trials who had received the investigational drug, olaparib in other research studies. There is no intervention given for this study.

This research is being done to understand of the mechanisms involved in patients whose cancer responds well and whose cancer does not respond well to investigational drug, olaparib, to help better understand how olaparib works and to better identify patients who may benefit from this therapy.

DETAILED DESCRIPTION:
This is study will compare biomarker research with response in patients who have received olaparib.

Patients who have had a durable response to olaparib for at least 2 years will be approached for the study.

Patients who agree to this study will then have their medical history collected and will be asked to complete a questionnaire. Archival tumor tissue will also be collected for biomarker research.

A waiver of consent is requested to access the medical records and archival tumor tissue of patients who are deceased.

If participants are still taking olaparib, they will be asked to provide blood samples for pharmacokinetics and circulating tumor DNA, and the results of CT scans taken as part of their standard of care or as a part of another research study. If participants' disease worsens while still on olaparib, they will then be asked to provide a blood sample for pharmacogenomics and BRCA testing (if not known). An optional tumor biopsy will also be requested.

Participants will continue to be followed by telephone for survival and any new treatments they are receiving.

ELIGIBILITY:
Inclusion Criteria:

* Previous or current treatment with Olaparib in a clinical trial/standard of care that included one of the following as a first step study for epithelial ovarian cancer (including fallopian tube or peritoneal cancer):

  * single agent olaparib given for relapsed disease or
  * single agent olaparib given as maintenance therapy after response to platinum based chemotherapy or
  * olaparib combined with platinum based chemotherapy and then continued as maintenance therapy or
  * olaparib combined with other types of therapy
* Had a durable response to Olaparib defined as patients who have benefited from olaparib for > 18 months. Patients who discontinued Olaparib due to toxicities but otherwise meet the definition of a durable response will be included or the control group is patients who had a short duration benefit with Olaparib of less than 6 months in any individual clinical trial/standard of care
* Ability to understand and the willingness to sign a written informed consent document.
* Patient's willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures.

Exclusion Criteria:

* Any severe acute or chronic medical or psychiatric condition or laboratory abnormality that would render the patient unsuitable for biopsy
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Epithelial ovarian cancer (including fallopian tube or peritoneal cancer) patients that are or had received treatment with Olaparib.
Sampling Method: Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
The number of patients with somatic BRCA mutations compared to number of patients without somatic BRCA mutations | 4 years
The number of patients with homologous recombination repair deficiencies compared to the number of patients that do not have homologous recombination repair deficiencies. | 4 years
The number and types of mutated genes. | 4 years
The number of patients with antibodies to the study drug | 4 years
Evaluate the levels of PI3K/Akt pathway expression per patient | 4 years

SECONDARY OUTCOMES:
HRR deficiency profile | 4 years
Level of poly (ADP-ribose) (PAR) expression | 4 years
Signature of PARP response compared with signature of platinum sensitivity | 4 years
Signature of PARP response and PARP resistance on different tumour sites | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (8):
- South Eastern Sydney Local Health District, Randwick, New South Wales, Australia
- Canada (3):
  - British Columbia Cancer Centre, Vancouver, British Columbia
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
- Institute of European Oncology, Milan, Italy
- Vall d'Hebron, Barcelona, Spain
- United Kingdom (2):
  - The Royal Marsden, Sutton, England
  - Edinburgh Cancer Research Centre, Edinburgh, Scotland